CLINICAL TRIAL: NCT03482856
Title: Cognitive Behavioural Therapy for Insomnia in Patients With Chronic Spinal Pain: a Multi-center Randomized Controlled Trial
Brief Title: Cognitive Behavioural Therapy for Insomnia in Chronic Spinal Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Vrije Universiteit Brussel (Other); Universitair Ziekenhuis Brussel (Other); University Hospital, Ghent (Other); Research Foundation Flanders (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EC/2018/0277
Record Dates: First submitted 2018-03-19; First posted 2018-03-29 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Chronic Low Back Pain; Chronic Neck Pain; Insomnia Chronic
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: The trial will randomize 120 patients with CSP and comorbid insomnia, aged between 18 and 65 years, to the experimental intervention (i.e. 18 sessions of the modern neuroscience approach combined with CBT-I, including 3 sessions of therapeutic pain neuroscience education, 6 sessions of CBT-I and 9 sessions of cognition-targeted exercise therapy, n=60) or the control intervention (i.e. 18 sessions of the modern neuroscience approach alone, including 3 sessions of therapeutic pain neuroscience education, and 15 sessions of cognition-targeted exercise therapy, n=60).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modern Neuroscience Approach (MNA) plus CBT-I (Experimental): MNA (i.e. modern pain neuroscience approach) combined with CBT-I (i.e. cognitive-behavioural therapy for insomnia)
  Interventions: Behavioral: MNA plus CBT-I
- MNA alone (Active Comparator): The MNA (i.e. modern pain neuroscience approach) alone
  Interventions: Behavioral: MNA alone

INTERVENTIONS:
Behavioral: MNA plus CBT-I — MNA plus CBT-I includes 3 sessions (1 group, 1 online and 1 individual session) of therapeutic pain neuroscience education, 6 individual sessions of CBT-I and 9 individual sessions of time-contingent dynamic and functional cognition-targeted exercise therapy, combined with home exercises. CBT-I is the standard evidence-based care for treating chronic primary insomnia and typically includes changing negative thoughts about sleep, sleep hygiene, sleep restriction therapy, and teaching relaxation skills. The 18 sessions will be spread over a period of 14 weeks.
  Arms: Modern Neuroscience Approach (MNA) plus CBT-I
Behavioral: MNA alone — MNA alone includes 3 sessions (1 group, 1 online and 1 individual session) of therapeutic pain neuroscience education, and 15 individual sessions of time-contingent dynamic and functional cognition-targeted exercise therapy, combined with home exercises. The 18 sessions will be spread over a period of 14 weeks.
  Arms: MNA alone

SUMMARY:
Chronic spinal pain (CSP) includes chronic low back and neck pain. CSP is a highly prevalent and severely debilitating disorder characterized by tremendous personal and socioeconomic impact, long-term sick leave, low quality of life and very high socioeconomical costs. The current strategies for treating CSP are not yet optimal in reducing pain and related disability, urging the need for improvement. A possible problem is that the current approaches are often to limited and only address pain.

Current treatments for CSP do not address associated complaints like sleeping problems which are however important issues. If present, sleeping problems may contribute to CSP severity and related disability. If left untreated, they represent a barrier for effective CSP management. Up to now, however, sleeping problems are hardly addressed and if so, it is mostly limited to sleeping medication. This is a problem since the efficacy and safety of drug treatment has not been established.

Therefore, within the current innovative project we propose examining the added value of cognitive behavioral therapy for insomnia (CBT-I) to the current best physical therapy treatment for CSP. CBT-I includes changing negative thoughts about sleep, sleep hygiene, altering sleeping patterns, and teaching relaxation skills.

The objectives of the study are to examine if CBT-I combined with the modern physical therapy approach (education about pain followed by exercise therapy) is more effective than the modern physical therapy approach alone for reducing pain, improving sleep and functionality in CSP patients with sleeping problems.

Therefore 120 CSP patients with sleeping problems will be randomly divided over the 2 treatment programs (60 per group) and will be assessed before and after their 14-week therapy program consisting of 18 therapy sessions. Comparisons will be made for pain severity, sleep quality and functionality.

DETAILED DESCRIPTION:
Modern pain neuroscience has advanced our understanding of chronic spinal pain (CSP). Despite the scientific progresses with regard to the treatment of chronic spinal pain (CSP), current treatments for CSP do not address pain comorbidities like insomnia, an important yet seldom addressed issue. Treatment of CSP mostly still relies on monotherapies or on biomedical models, as shown by expensive but ineffective treatments like lumbar fusion surgery, ignoring important comorbidities such as insomnia.

Within the current innovative project we propose examining the added value of cognitive behavioral therapy for insomnia (CBT-I) to the current best evidence treatment for CSP. The innovative nature of this approach to CSP goes well beyond the combination of 2 available and effective treatments: combining cognitive behavioral therapy for insomnia with the recently established modern neuroscience approach (pain neuroscience education followed by cognition-targeted exercise therapy) strengthens the content of both individual approaches and applies the current understanding regarding insomnia and pain neuroscience to clinical practice. This innovative combination will result in a synergistic effect of both treatments.

The primary scientific objective of the study is to examine if CBT-I combined with a modern neuroscience approach (pain neuroscience education followed by cognition-targeted exercise therapy) is more effective than the modern neuroscience approach alone for reducing pain in CSP patients with insomnia. Secondary objectives of the study are to examine if CBT-I combined with the modern neuroscience approach is more effective than the modern neuroscience approach alone for improving pain related outcomes, sleep related outcomes and physical activity/functionality in CSP patients with insomnia.

To comply with these scientific objectives, the 120 CSP patients with comorbid insomnia will be subjected to the baseline assessment of all outcome measures.

Follow-up assessments will be performed immediately after 14 weeks of therapy (all tests), and 3 months (questionnaires), 6 months (questionnaires) and 12 months (all tests, depending on a go/no go decision) after finishing the therapeutic intervention.

To investigate these objectives, a muli-center triple-blind randomized, controlled trial with 1 year follow up will be performed.

Appropriate statistical analyses will be performed to evaluate and compare treatment effects. Statistical, as well as clinical significant differences will be defined and the effect size will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Nonspecific spinal pain for at least 3 months' duration, at least 3 days per week
* Seeking care because of neck pain or low back pain
* Native Dutch speaker
* Having insomnia: in the absence of other intrinsic sleep disorders and shift work, insomnia is defined as > 30 minutes of sleep latency and/or minutes awake after sleep onset for > 3 days / week for > 6 months
* Living or working within a radius of 50 km around the therapy location
* Not starting new treatments or medication and continuing their usual care 6 weeks prior to and during study participation (to obtain a steady state)
* Refraining from analgesics, caffeine, alcohol or nicotine in the previous 48h of the assessments
* Nonspecific failed back surgery > 3 years are permitted
* Not undertaking exercise (> 3 metabolic Equivalents) 3 days before the assessments

Exclusion Criteria:

* Severe underlying sleep pathology (identified through baseline data of polysomnography)
* Neuropathic pain
* Chronic widespread pain
* Being pregnant or pregnancy (including given birth) in the preceding year
* History of specific spinal surgery
* Thoracic pain in absence of neck or low back pain
* Shift workers
* Diagnosed depression
* Body Mass Index below 30

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Brief Pain Inventory (Numeric Rating Scale) | Baseline assessment, T1 follow-up assessment after 14 weeks of therapy, T2 follow-up assessment 3 months after the end of therapy, T3 follow-up assessment 6 months after the end of therapy, and T4 follow-up assessment 12 months after the end of therapy
  Change in self-reported pain: The question "please rate your pain by circling the one number that best describes your pain on the AVERAGE" is used as the primary outcome measure to evaluate pain intensity. Scale ranges from 0 to 10, with higher scores indicating more self-reported pain.

SECONDARY OUTCOMES:
Brief Pain Inventory | Baseline assessment, T1 follow-up assessment after 14 weeks of therapy, T2 follow-up assessment 3 months after the end of therapy, T3 follow-up assessment 6 months after the end of therapy, and T4 follow-up assessment 12 months after the end of therapy
  Change in self-reported impact of pain on functioning. Scale ranges from 0 to 10, with higher scores indicating more self-reported pain or higher interference of pain in daily life.
Central Sensitization Inventory | Baseline assessment, T1 follow-up assessment after 14 weeks of therapy, T2 follow-up assessment 3 months after the end of therapy, T3 follow-up assessment 6 months after the end of therapy, and T4 follow-up assessment 12 months after the end of therapy
  Change in self-reported central sensitization symptoms. Score ranges from 0 to 100, with higher scores indicating more self-reported symptoms of central sensitization.
Pressure Pain Thresholds | Baseline assessment, T1 follow-up assessment after 14 weeks of therapy, and T4 follow-up assessment 12 months after the end of therapy
  Change in Pressure Pain Thresholds at measured bilaterally with a digital pressure algometer (Wagner Instruments), both at symptomatic levels (trapezius muscle and 5 centimetres lateral to the spinous process of L3) and at remote sites (i.e. secondary hyperalgesia).
Polysomnography (PSG) | Baseline assessment, T1 follow-up assessment after 14 weeks of therapy, and T4 follow-up 12 months after the end of therapy. Polysomnography T4 assessment will be carried out based on a go/no go decision, if improvements are visible at the T1 assessment.
  Change in polysomnography. Participants will be monitored in the comfort of their own home by ambulatory PSG.
Pittsburg Sleep Quality Index | Baseline assessment, T1 follow-up assessment after 14 weeks of therapy, T2 follow-up assessment 3 months after the end of therapy, T3 follow-up assessment 6 months after the end of therapy, and T4 follow-up assessment 12 months after the end of therapy
  Change in self-reported perceived sleep quality. Score ranges from 0 to 21, 0 indicating no difficulty and 21 indicating severe sleep difficulties.
Insomnia Severity Index | Baseline assessment, T1 follow-up assessment after 14 weeks of therapy, T2 follow-up assessment 3 months after the end of therapy, T3 follow-up assessment 6 months after the end of therapy, and T4 follow-up assessment 12 months after the end of therapy
  Change in self-reported insomnia severity. Score ranges from 0 to 28, with 0 indicating no clinically significant insomnia and 28 indicating severe clinical insomnia.
DBAS (i.e. Dysfunctional Beliefs and Attitudes about Sleep) | Baseline assessment, T1 follow-up assessment after 14 weeks of therapy, T2 follow-up assessment 3 months after the end of therapy, T3 follow-up assessment 6 months after the end of therapy, and T4 follow-up assessment 12 months after the end of therapy
  Change in self-reported dysfunctional beliefs and attitudes about sleep. Score ranges from 0 to 10. Scores above 4 indicate unrealistic expectations for sleep or unrealistic thoughts about sleep.
Epworth Sleepiness Scale | Baseline assessment, T1 follow-up assessment after 14 weeks of therapy, T2 follow-up assessment 3 months after the end of therapy, T3 follow-up assessment 6 months after the end of therapy, and T4 follow-up assessment 12 months after the end of therapy
  Change in self-reported sleep propensity. Score ranges from 0 to 24, with 0 indicating normal daytime sleepiness and 24 indicating severe excessive daytime sleepiness.
Brugmann Fatigue Scale | Baseline assessment, T1 follow-up assessment after 14 weeks of therapy, T2 follow-up assessment 3 months after the end of therapy, T3 follow-up assessment 6 months after the end of therapy, and T4 follow-up assessment 12 months after the end of therapy
  Change in self-reported fatigue severity. Score ranges from 0 to 24, with higher scores indicating higher subjective levels of fatigue.
Hospital Anxiety and Depression rating scale | Baseline assessment, T1 follow-up assessment after 14 weeks of therapy, T2 follow-up assessment 3 months after the end of therapy, T3 follow-up assessment 6 months after the end of therapy, and T4 follow-up assessment 12 months after the end of therapy
  Change in self-reported affective symptoms. Score ranges from 0 to 21, with 0 indicating absence of depression or anxiety and 21 indicating the presence of depression or anxiety.
Physical Activity using Actigraphy | 1 week at baseline, 1 week at T1 follow-up assessment after 14 weeks of therapy, 1 week at T4 follow-up assessment 12 months after the end of therapy
  Change in physical activity: Continuous assessment of physical activity and rest/activity cycles
Short Form Health Survey - 36 items Mental Health | Baseline assessment, T1 follow-up assessment after 14 weeks of therapy, T2 follow-up assessment 3 months after the end of therapy, T3 follow-up assessment 6 months after the end of therapy, and T4 follow-up assessment 12 months after the end of therapy
  Change in self-reported functional status and well-being or quality of life. Score ranges from 0 to 400 with higher scores indicating better mental health.
Short Form Health Survey - 36 items Physical Health | Baseline assessment, T1 follow-up assessment after 14 weeks of therapy, T2 follow-up assessment 3 months after the end of therapy, T3 follow-up assessment 6 months after the end of therapy, and T4 follow-up assessment 12 months after the end of therapy
  Change in self-reported functional status and well-being or quality of life. Score ranges from 0 to 400 with higher scores indicating better physical health.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Cagnie, PhD, Principal Investigator — University Ghent
Locations (2):
- Belgium (2):
  - University Hospital Brussels, Brussels, Brussels Capital
  - University Hospital Ghent, Ghent, Oost-Vlaanderen

REFERENCES:
- [Background] Nijs J, Meeus M, Cagnie B, Roussel NA, Dolphens M, Van Oosterwijck J, Danneels L. A modern neuroscience approach to chronic spinal pain: combining pain neuroscience education with cognition-targeted motor control training. Phys Ther. 2014 May;94(5):730-8. doi: 10.2522/ptj.20130258. Epub 2014 Jan 30. PMID 24481595
- [Background] Nijs J, Mairesse O, Neu D, Leysen L, Danneels L, Cagnie B, Meeus M, Moens M, Ickmans K, Goubert D. Sleep Disturbances in Chronic Pain: Neurobiology, Assessment, and Treatment in Physical Therapist Practice. Phys Ther. 2018 May 1;98(5):325-335. doi: 10.1093/ptj/pzy020. PMID 29425327
- [Background] Nijs J, Lluch Girbes E, Lundberg M, Malfliet A, Sterling M. Exercise therapy for chronic musculoskeletal pain: Innovation by altering pain memories. Man Ther. 2015 Feb;20(1):216-20. doi: 10.1016/j.math.2014.07.004. Epub 2014 Jul 18. PMID 25090974
- [Background] Malfliet A, Kregel J, Meeus M, Cagnie B, Roussel N, Dolphens M, Danneels L, Nijs J. Applying contemporary neuroscience in exercise interventions for chronic spinal pain: treatment protocol. Braz J Phys Ther. 2017 Sep-Oct;21(5):378-387. doi: 10.1016/j.bjpt.2017.06.019. Epub 2017 Jul 8. PMID 28736211
- [Derived] Malfliet A, De Baets L, Bilterys T, Van Looveren E, Mairesse O, Cagnie B, Meeus M, Moens M, Goubert D, Munneke W, Daneels L, Ickmans K, Kamper S, Nijs J. Cognitive Behavioral Therapy for Insomnia in Pain Management for Nonspecific Chronic Spinal Pain: A Randomized Clinical Trial. JAMA Netw Open. 2024 Aug 1;7(8):e2425856. doi: 10.1001/jamanetworkopen.2024.25856. PMID 39120902
- [Derived] Malfliet A, Bilterys T, Van Looveren E, Meeus M, Danneels L, Ickmans K, Cagnie B, Mairesse O, Neu D, Moens M, Goubert D, Kamper SJ, Nijs J. The added value of cognitive behavioral therapy for insomnia to current best evidence physical therapy for chronic spinal pain: protocol of a randomized controlled clinical trial. Braz J Phys Ther. 2019 Jan-Feb;23(1):62-70. doi: 10.1016/j.bjpt.2018.10.007. Epub 2018 Oct 29. PMID 30389347